CLINICAL TRIAL: NCT02635815
Title: Risk Factors for Variceal Bleeding in Egyptian Patients With Non-Cirrhotic Portal Hypertension
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Abdelhakam, Assistant Professor, Ain Shams University
Other Study IDs: 699
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group I: twenty six patients with history of bleeding or had an attack of bleeding during one year follow-up. All underwent upper gastrointestinal endoscopy.
  Interventions: Procedure: Upper gastrointestinal endoscopy
- Group II: thirty four patients without bleeding. All underwent upper gastrointestinal endoscopy.
  Interventions: Procedure: Upper gastrointestinal endoscopy

INTERVENTIONS:
Procedure: Upper gastrointestinal endoscopy — Upper gastrointestinal endoscopy using the Pentax video endoscope EG 3440

SUMMARY:
Background & Aims: Non-cirrhotic portal hypertension (NCPH) represents a relatively infrequent group of conditions. This work aimed at determining causes of NCPH and evaluating the role of some clinical, laboratory, imaging and endoscopic parameters in prediction of variceal bleeding in an Egyptian cohort with NCPH.

Methods: Sixty patients with non-cirrhotic portal hypertension and oesophageal varices were included. All underwent complete clinical evaluation, laboratory investigations, Color Doppler ultrasonography, platelet count/spleen diameter (mm) ratio and upper gastrointestinal endoscopy. Patients were classified into two groups according to variceal bleeding: (1) Group I: twenty six patients with history of bleeding or had an attack of bleeding during one year follow-up; and (2) Group II: thirty four patients without bleeding.

DETAILED DESCRIPTION:
All of the included patients underwent: (1) A complete clinical evaluation; (2) Laboratory investigations: CBC, liver profile, viral markers (HBs Ag, HB core Ab, HCV Ab) using the ELISA technique; (3) Thrombophilia workup to clarify the underlying etiology of vascular liver disease. It was done only for patients with Budd-Chiari syndrome and extrahepatic portal vein thrombosis: anticardiolipin antibodies, lupus anticoagulant, antinuclear antibodies, protein C, S, antithrombin III, factor V Leiden G1691A mutation, prothrombin gene G20210A mutation, methylene tetrahydrofolate reductase C677T mutation by PCR, Janus tyrosine kinase-2 (JAK II) V617F mutation by PCR (to exclude myeloproliferative disorders) and flow cytometry for CD55 and CD59 (to exclude paroxysmal nocturnal hemoglobinuria); (4) Abdominal ultrasonography: for liver size, echogenicity, spleen size, portal vein diameter and ascites; (5) Color Doppler ultrasonographic study: was done in the morning after an overnight fasting using a color Doppler unit with a 3.5 MHz convex probe for confirmation of portal vein (PV) patency and diameter, mean PV flow velocity (mean PVV) (cm/sec), PV direction of flow, splenic vein patency and diameter, presence of portosystemic collaterals and patency of hepatic veins; (6) Platelet count/spleen diameter ratio: calculated as: platelet count/ maximum spleen bipolar diameter by ultrasound in mm; (7) Ultrasonography guided liver biopsy: for diagnosis of NCPH and exclusion of cirrhotic portal hypertension; and (8) Upper gastrointestinal endoscopy using the Pentax video endoscope EG 3440. Oesophageal varices were classified according to their size into small, medium or large [8]. Prophylaxis with band ligation was done to patients with large or medium sized risky varices who were eligible for starting anticoagulation. The diagnosis of variceal bleeding was confirmed if an actively bleeding varix or a varix with adherent clot or white nipple was seen. Red color signs were classified into Cherry Red Spots "CRS", Red Wale Markings "RWM" and Hematocystic Spots "HCS". Gastric varices were classified into either gastro-esophageal varices (GEV) or isolated gastric varices (IGV). Portal hypertensive gastropathy (PHG) was classified into either mild or severe.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian patients with non-cirrhotic portal hypertension (NCPH) with oesophageal varices

Exclusion Criteria:

* Patients with concomitant infection with viral hepatitis, cirrhotic portal hypertension, hepatocellular carcinoma as well as those with other sources of bleeding such as erosions or ulcers were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian patients with non-cirrhotic portal hypertension (NCPH) with oesophageal varices, presenting with or without variceal bleeding
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The presence or absence of variceal bleeding within one year of follow up. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Reda Elwakil, Professor, Study Director — Ain Shams University